CLINICAL TRIAL: NCT05975606
Title: Exploring the Effect of Non-invasive Brain Stimulation Paired With Functional Electrical Stimulation to Improve Lower Extremity Function Following Incomplete Spinal Cord Injury
Brief Title: Non-invasive Brain Stimulation Paired With FES Cycling Post SCI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Western University, Canada (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 122650
Record Dates: First submitted 2023-07-10; First posted 2023-08-04 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2024-07

CONDITIONS: Incomplete Spinal Cord Injury
Keywords: incomplete spinal cord injury; repetitive transcranial magnetic stimulation; functional electrical stimulation cycling; lower extremity function; walking speed; muscle strength; feasibility
MeSH Terms: interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: This protocol involves two groups of participants: intervention group and control group. Intervention group will receive real rTMS and FES cycling and control group will receive sham rTMS and FES cycling. The results of these groups are then evaluated at several stages of the study.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Participants are blinded to their groups. Research assistant and physiotherapist who are responsible for conducting assessment sessions are also blinded to participants group.
  All the participants will be randomized to groups using opaque envelopes blocked by four and stratified by AIS score.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment group (Experimental): Participants of this group will receive active rTMS along with real FES cycling.
  Interventions: Device: repetitive transcranial magnetic stimulation (rTMS); Device: functional electrical stimulation (FES) cycling
- Control group (Sham Comparator): Participants of this group will receive sham rTMS along with real FES cycling.
  Interventions: Device: functional electrical stimulation (FES) cycling

INTERVENTIONS:
Device: repetitive transcranial magnetic stimulation (rTMS) — rTMS will be applied to primary motor cortex of the brain.
  Arms: Treatment group
Device: functional electrical stimulation (FES) cycling — FES will be applied to muscles associated in cycling: quadriceps, hamstrings, tibialis anterior, gastrocnemius, soleus.

SUMMARY:
This project is randomized controlled trial which will explore the effect of pairing repetitive Transcranial Magnetic Stimulation (rTMS) with Functional Electrical Stimulation (FES) Cycling on lower extremity function in people with incomplete spinal cord injury and compare the effects to each one of these interventions alone.

DETAILED DESCRIPTION:
Following a spinal cord injury, people often have decreased strength and balance in their legs, making it difficult to walk. To improve leg function in people with spinal cold injuries, the investigators can use electrical stimulation on muscles while participants are cycling to increase the muscle activation and nerve connections. Another way to improve the nerve connections to the muscles is by stimulating the brain directly. Previous research has looked at the effects of each of these treatments, but they have not been used together. In this study, the investigators will pair both electrical stimulation on the legs during cycling with brain stimulation or a sham brain stimulation to improve recovery and determine if using these methods together results in better outcomes, such as increased walking speed. Participants will attend training sessions for six weeks, twice per week. Each person will first receive the active or sham brain stimulation at the beginning of the session for 30 minutes and then they will receive the electrical stimulation on their legs while cycling for 60 minutes. Participants will be evaluated before the start of the treatment, in the middle of the study, at the final session, and again two weeks after the last session of the treatment. Assessments will include clinical tests of gait, balance, and strength. Inertial Measurement Units (IMU) and a pressure sensor gait mat will be used to evaluate the gait and balance parameters.

ELIGIBILITY:
Inclusion Criteria:

* adult
* having motor incomplete SCI with level C or D on the American Spinal Injury Association Impairment Scale (AIS) with the lesion at any level of the cord resulting from either traumatic or non-traumatic etiology who are at least one-year post-injury.
* having non-progressive SCI
* being able to walk independently for 10 meters without help from another person

Exclusion Criteria:

* other orthopedic or neurological implications that affect the lower extremity function
* contraindications to FES (e.g., implanted electronic devices, unhealed bone fractures, sever contractures, extreme osteoporosis or osteoarthritis)
* contraindications to rTMS (e.g., metal implants, history of seizure, cochlear implants)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2023-09-19 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Time taken to complete the recruitment of 12 participants | 8 weeks
  This outcome will be evaluated through descriptive data. This outcome will be analyzed to evaluate the feasibility of the protocol.
Proportion of participants recruited from the total number screened | 8 weeks
  This outcome will be evaluated through descriptive data. This outcome will be analyzed to evaluate the feasibility of the protocol.
Number of sessions attended by each participant | 8 weeks
  This outcome will be evaluated through descriptive data. This outcome will be analyzed to evaluate the tolerability of the protocol.
Number of dropouts in each group | 8 weeks
  This outcome will be evaluated through descriptive data. This outcome will be analyzed to evaluate the tolerability of the protocol.
Willingness of participants to undergo therapy | 8 weeks
  This outcome will be evaluated through descriptive data. This outcome will be analyzed to evaluate the tolerability of the protocol. The willingness of participation will be collected on an 11-point numerical rating scale with 'not at all willing' at 0, and 'very willing' at 10 (measured at baseline).
Incidence of treatment-emergent adverse events | 8 weeks
  This outcome will be evaluated through descriptive data. Safety will be presented as any adverse reaction reported on verbal questioning at each session. The number of participants reporting adverse reactions, and the duration and severity of the adverse reactions will be reported.

SECONDARY OUTCOMES:
Walking speed | 8 weeks
  This instrumental outcome is collected using a pressure sensor gait mat.
Step length | 8 weeks
  This instrumental outcome is collected using a pressure sensor gait mat.
Step width | 8 weeks
  This instrumental outcome is collected using a pressure sensor gait mat.
Cadence | 8 weeks
  This instrumental outcome is collected using a pressure sensor gait mat.
Timed Up and Go (TUG) test | 8 weeks
  This instrumental outcome will be collected using Inertial Measurement Units (IMUs).
Sit-to-stand test | 8 weeks
  This instrumental outcome will be collected using Inertial Measurement Units (IMUs).
Postural sway test | 8 weeks
  This instrumental outcome will be collected using Inertial Measurement Units (IMUs).
Lower Extremity Motor Score (LEMS) | 8 weeks
  A blinded physiotherapist will be hired to collect this clinical outcome.
  Lower Extremity Motor Score is rated from 0 to 5* as follows:
  0= Total paralysis
  1. Palpable or visible contraction
  2. Active movement, full range of motion (ROM) when gravity is eliminated
  3. Active movement, full ROM against gravity
  4. Active movement, full ROM against gravity, and moderate resistance in muscle-specific position
  5. (Normal) Active movement, full ROM against gravity, and full resistance in a muscle-specific position expected from a healthy person 5*= (Normal) Active movement, full ROM against gravity, and sufficient resistance to be considered normal if identified inhibiting factors (i.e., pain, disuse) were not present NT = Not testable (i.e., due to immobilization, sever pain that can prevent the grading of the patient, amputation of the limb, or contracture of >50% of the range of motion) Higher scores in this outcome mean better result.
Walking Index for Spinal Cord Injury (WISCI) II scale | 8 weeks
  A blinded physiotherapist will be hired to collect this clinical outcome. Walking Index for Spinal Cord Injury version II scale is rated from 0 to 20 with the higher scores showing better results.

OTHER OUTCOMES:
Global Rating of Change (GRC) scale | 8 weeks
  Evaluation of the participants' impact will be collected through a GRC questionnaire in each assessment session.
  Global Rating Scale will ask participants to rate their walking abilities and overall recovery of the lower limb function from the time that they began the treatment until now. This scale is rated from -7 to 7 as follows:
  * 7: A very great deal worse
  * 6: A great deal worse
  * 5: Quite a bit worse
  * 4: Moderately worse
  * 3: Somewhat worse
  * 2: A little bit worse
  * 1: A tiny bit worse (almost the same) 0: About the same
    * 1: A tiny bit better (almost the same)
    * 2: A little bit better
    * 3: Somewhat better
    * 4: Moderately better
    * 5: Quite a bit better
    * 6: A great deal better
    * 7: A very great deal better
  Higher scores in this outcome mean better results.

CONTACTS AND LOCATIONS:
Overall Officials: Siobhan Schabrun, PhD, Study Director — Western University, Canada
Locations (1):
- Parkwood Institute, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
IPD of this study will not be shared with other researchers of other studies.

REFERENCES:
- [Background] Ding W, Hu S, Wang P, Kang H, Peng R, Dong Y, Li F. Spinal Cord Injury: The Global Incidence, Prevalence, and Disability From the Global Burden of Disease Study 2019. Spine (Phila Pa 1976). 2022 Nov 1;47(21):1532-1540. doi: 10.1097/BRS.0000000000004417. Epub 2022 Jun 30. PMID 35857624
- [Background] Qin W, Bauman WA, Cardozo C. Bone and muscle loss after spinal cord injury: organ interactions. Ann N Y Acad Sci. 2010 Nov;1211:66-84. doi: 10.1111/j.1749-6632.2010.05806.x. PMID 21062296
- [Background] REED WB, PIDGEON J, BECKER SW. Patients with spinal cord injury. Clinical cutaneous studies. Arch Dermatol. 1961 Mar;83:379-85. doi: 10.1001/archderm.1961.01580090029002. No abstract available. PMID 13740272
- [Background] Riggins MS, Kankipati P, Oyster ML, Cooper RA, Boninger ML. The relationship between quality of life and change in mobility 1 year postinjury in individuals with spinal cord injury. Arch Phys Med Rehabil. 2011 Jul;92(7):1027-33. doi: 10.1016/j.apmr.2011.02.010. PMID 21704781
- [Background] Sadowsky CL, Hammond ER, Strohl AB, Commean PK, Eby SA, Damiano DL, Wingert JR, Bae KT, McDonald JW 3rd. Lower extremity functional electrical stimulation cycling promotes physical and functional recovery in chronic spinal cord injury. J Spinal Cord Med. 2013 Nov;36(6):623-31. doi: 10.1179/2045772313Y.0000000101. Epub 2013 Mar 20. PMID 24094120
- [Background] BARRIA P, AGUILAR R, DS D, MORIS A, ANDRADE A, JM A. Instrumented gait analysis of stroke patients after FES-cycling therapy.
- [Background] Benito J, Kumru H, Murillo N, Costa U, Medina J, Tormos JM, Pascual-Leone A, Vidal J. Motor and gait improvement in patients with incomplete spinal cord injury induced by high-frequency repetitive transcranial magnetic stimulation. Top Spinal Cord Inj Rehabil. 2012 Spring;18(2):106-12. doi: 10.1310/sci1802-106. PMID 23459246
- [Background] Fawaz S, Kamel F, El Yasaky A, El Shishtawy H, Genedy A, Awad RM, El Nabil L. The therapeutic application of functional electrical stimulation and transcranial magnetic stimulation in rehabilitation of the hand function in incomplete cervical spinal cord injury. Egyptian Rheumatology and Rehabilitation. 2019 Jan;46(1):21-6.
- [Background] Shariat A, Hosseini L, Najafabadi MG, Cleland JA, Shaw BS, Shaw I. Functional Electrical Stimulation and Repetitive Transcranial Magnetic Stimulation for Neurorehabilitation in Patients Post Stroke: A Short Communication. Asian Journal of Sports Medicine. 2018 Dec 31;9(4).
- [Background] Krogh S, Aagaard P, Jonsson AB, Figlewski K, Kasch H. Effects of repetitive transcranial magnetic stimulation on recovery in lower limb muscle strength and gait function following spinal cord injury: a randomized controlled trial. Spinal Cord. 2022 Feb;60(2):135-141. doi: 10.1038/s41393-021-00703-8. Epub 2021 Sep 9. PMID 34504284
- [Background] Alexeeva N, Calancie B. Efficacy of QuadroPulse rTMS for improving motor function after spinal cord injury: Three case studies. J Spinal Cord Med. 2016;39(1):50-7. doi: 10.1179/2045772314Y.0000000279. Epub 2014 Dec 1. PMID 25437531
- [Background] Kumru H, Benito J, Murillo N, Valls-Sole J, Valles M, Lopez-Blazquez R, Costa U, Tormos JM, Pascual-Leone A, Vidal J. Effects of high-frequency repetitive transcranial magnetic stimulation on motor and gait improvement in incomplete spinal cord injury patients. Neurorehabil Neural Repair. 2013 Jun;27(5):421-9. doi: 10.1177/1545968312471901. Epub 2013 Jan 15. PMID 23322551
- [Background] Kumru H, Benito-Penalva J, Valls-Sole J, Murillo N, Tormos JM, Flores C, Vidal J. Placebo-controlled study of rTMS combined with Lokomat(R) gait training for treatment in subjects with motor incomplete spinal cord injury. Exp Brain Res. 2016 Dec;234(12):3447-3455. doi: 10.1007/s00221-016-4739-9. Epub 2016 Jul 28. PMID 27469242
- [Background] Donaldson N, Perkins TA, Fitzwater R, Wood DE, Middleton F. FES cycling may promote recovery of leg function after incomplete spinal cord injury. Spinal Cord. 2000 Nov;38(11):680-2. doi: 10.1038/sj.sc.3101072. PMID 11114775
- [Background] Sloan KE, Bremner LA, Byrne J, Day RE, Scull ER. Musculoskeletal effects of an electrical stimulation induced cycling programme in the spinal injured. Paraplegia. 1994 Jun;32(6):407-15. doi: 10.1038/sc.1994.67. PMID 8090549
- [Background] Mazzoleni S, Stampacchia G, Gerini A, Tombini T, Carrozza MC. FES-cycling training in spinal cord injured patients. Annu Int Conf IEEE Eng Med Biol Soc. 2013;2013:5339-41. doi: 10.1109/EMBC.2013.6610755. PMID 24110942
- [Background] Waters RL, Adkins RH, Yakura JS, Sie I. Motor and sensory recovery following incomplete paraplegia. Arch Phys Med Rehabil. 1994 Jan;75(1):67-72. PMID 8291966
- [Background] Wang RY, Wang FY, Huang SF, Yang YR. High-frequency repetitive transcranial magnetic stimulation enhanced treadmill training effects on gait performance in individuals with chronic stroke: A double-blinded randomized controlled pilot trial. Gait Posture. 2019 Feb;68:382-387. doi: 10.1016/j.gaitpost.2018.12.023. Epub 2018 Dec 18. PMID 30586670
- [Background] Shariat A, Najafabadi MG, Ansari NN, Cleland JA, Singh MAF, Memari AH, Honarpishe R, Hakakzadeh A, Ghaffari MS, Naghdi S. The effects of cycling with and without functional electrical stimulation on lower limb dysfunction in patients post-stroke: A systematic review with meta-analysis. NeuroRehabilitation. 2019;44(3):389-412. doi: 10.3233/NRE-182671. PMID 31227660